CLINICAL TRIAL: NCT03462706
Title: A Randomized Trial Comparing the Effectiveness of Polyp Resection Treatments (Hot Snare vs Cold Snare vs Hot EMR vs Cold EMR)
Brief Title: Quad Resection (Hot Snare vs Cold Snare vs Hot EMR vs Cold EMR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: John D. Dingell VA Medical Center (U.S. Federal Agency); White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Douglas K. Rex, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1711062130
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Colon Cancer; Colon Polyp; Colon Adenoma
Keywords: Polyp Resection; Cold Snare; Hot Snare; Cold Endoscopic Mucosal Resection (EMR); Hot Endoscopic Mucosal Resection (EMR); Colonoscopy
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold Snare (Experimental): Polyps sized 6mm to 15mm found during colonoscopy will be removed using cold snare techniques.
  Interventions: Procedure: Cold Snare
- Hot Snare (Experimental): Polyps sized 6mm to 15mm found during colonoscopy will be removed using hot snare techniques.
  Interventions: Procedure: Hot Snare
- Cold EMR (Experimental): Polyps sized 6mm to 15mm found during colonoscopy will be removed using cold EMR techniques.
  Interventions: Procedure: Cold EMR
- Hot EMR (Experimental): Polyps sized 6mm to 15mm found during colonoscopy will be removed using hot EMR techniques.
  Interventions: Procedure: Hot EMR

INTERVENTIONS:
Procedure: Cold Snare — Subjects randomized to Cold Snare Intervention will have any polyps sized 6mm to 15mm removed using cold snare techniques (no electrocautery, no submucosal injection.)
  Arms: Cold Snare
Procedure: Hot Snare — Subjects randomized to Hot Snare Intervention will have any polyps sized 6mm to 15mm removed using hot snare techniques (with electrocautery, no submucosal injection.)
  Arms: Hot Snare
Procedure: Cold EMR — Subjects randomized to Cold EMR will have any polyps sized 6mm to 15mm removed using cold EMR techniques (no electrocautery, with submucosal injection.)
  Arms: Cold EMR
Procedure: Hot EMR — Subjects randomized to Hot EMR will have any polyps sized 6mm to 15mm removed using hot EMR techniques (with electrocautery, with submucosal injection.)
  Arms: Hot EMR

SUMMARY:
The study will compare the use of cold snare, hot snare, cold EMR, and hot EMR for polyp resection. Although previous studies have compared two of the potential resection methods, no previous study has evaluated all four of the resection methods.

DETAILED DESCRIPTION:
The optimal method for removal of polyps 6-9 and 10-15 mm in size is not established. In this study, we propose to evaluate four different treatments for polyps (sized 6mm-15mm). The four treatments are cold snaring without injection, hot snaring without injection, cold EMR, and hot EMR. This study aims to help to establish the optimal resection technique for 6-9 and 10-15 mm polyps.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older
* Ability to provide informed consent

Exclusion Criteria:

* Subjects with a history of Inflammatory Bowel Disease
* Lesions less than 6mm or greater than 15mm in largest dimension

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared in the future upon request per PI discretion.

REFERENCES:
- [Derived] Rex DK, Anderson JC, Pohl H, Lahr RE, Judd S, Antaki F, Lilley K, Castelluccio PF, Vemulapalli KC. Cold versus hot snare resection with or without submucosal injection of 6- to 15-mm colorectal polyps: a randomized controlled trial. Gastrointest Endosc. 2022 Aug;96(2):330-338. doi: 10.1016/j.gie.2022.03.006. Epub 2022 Mar 12. PMID 35288147

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cold Snare | Cold EMR | Hot Snare | Hot EMR
Started | 60 | 63 | 58 | 57
Completed | 59 | 63 | 57 | 56
Not Completed | 1 | 0 | 1 | 1
Not completed — Polyp was pedunculated | 1 | 0 | 1 | 0
Not completed — Polyp was next to a cancer and not removed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cold Snare | Cold EMR | Hot Snare | Hot EMR | Total
Number analyzed (Participants) | 59 | 63 | 57 | 56 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (9.9) | 65.0 (8.0) | 66.3 (8.0) | 67.0 (8.4) | 66.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 19 | 17 | 89
  Male | 34 | 35 | 38 | 39 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 2 | 1 | 6 | 11
  White | 56 | 60 | 54 | 48 | 218
  Other/Unknown | 1 | 1 | 2 | 2 | 6
Number of Polyps [Number; unit: Polyps] | 68 | 82 | 71 | 65 | 286
Indication [Count of Participants; unit: Participants]
  Diagnostic | 7 | 7 | 4 | 6 | 24
  Screening | 17 | 10 | 8 | 8 | 43
  Surveillance | 34 | 43 | 40 | 41 | 158
  Therapeutic | 1 | 3 | 5 | 1 | 10
Site [Count of Participants; unit: Participants]
  Indiana University | 44 | 47 | 41 | 37 | 169
  Detroit Veterans Affairs Medical Center | 6 | 2 | 4 | 9 | 21
  White River Junction Veterans Affairs Medical Center | 9 | 14 | 12 | 10 | 45

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Resection (Central Post-Resection Biopsies)
Description: Efficacy of resection will be assessed by biopsies in four quadrants of the perimeter of the defect post-resection and one biopsy from the center of the defect post-resection. Comparison of the biopsy pathology results for polyps removed by cold snare vs. hot snare vs. cold EMR vs. hot EMR. Negative means that there was no residual polyp tissue seen on the central post-resection biopsies. Positive means that there was residual polyp tissue seen on the central post-resection biopsies. Negative central post-resection biopsies are considered a better outcome.
Time Frame: 1 day
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Cold Snare | Cold EMR | Hot Snare | Hot EMR
Number analyzed (Participants) | 59 | 63 | 57 | 56
Number analyzed (Polyps) | 68 | 82 | 71 | 65
Polyps
  Negative | 68 | 82 | 69 | 63
  Positive | 0 | 0 | 2 | 2

2. Primary Outcome: Efficacy of Resection (Peripheral Post-Resection Biopsies)
Description: Efficacy of resection will be assessed by biopsies in four quadrants of the perimeter of the defect post-resection and one biopsy from the center of the defect post-resection. Comparison of the biopsy pathology results for polyps removed by cold snare vs. hot snare vs. cold EMR vs. hot EMR. Negative means that there was no residual polyp tissue seen on the peripheral post-resection biopsies. Positive means that there was residual polyp tissue seen on the peripheral post-resection biopsies. Negative peripheral post-resection biopsies are considered a better outcome.
Time Frame: 1 day
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Cold Snare | Cold EMR | Hot Snare | Hot EMR
Number analyzed (Participants) | 59 | 63 | 57 | 56
Number analyzed (Polyps) | 68 | 82 | 71 | 65
Polyps
  Negative | 68 | 81 | 70 | 62
  Positive | 0 | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: 1 month
Description: Patients were called approximately 30 days after their colonoscopy procedure.
Arm/Group | Cold Snare | Cold EMR | Hot Snare | Hot EMR
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/63 | 0/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/63 | 1/57 | 1/56
Other Adverse Events (participants affected / at risk) | 8/59 | 11/63 | 10/57 | 6/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cold Snare (N=59) | Cold EMR (N=63) | Hot Snare (N=57) | Hot EMR (N=56)
delayed hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Delayed bleeding requiring treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cold Snare (N=59) | Cold EMR (N=63) | Hot Snare (N=57) | Hot EMR (N=56)
Intraprocedural bleed from biopsy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Delayed Bleed (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 2 (2) | 1 (1) — Bleeding noticed after procedure but not requiring intervention
Abdominal pain (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 2 (2) | 1 (1)
Urinary incontinence or retention (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bowel Movement Irregularity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Medication Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Other, Miscellaneous (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study endoscopists are experts with special interest in polypectomy; serrated lesions were included in the study instead of only including adenomas; incomplete resections occurred in 10-15mm lesions so a study designed for 10-15mm or 10-20mm lesions may be more relevant; potential of proceduralist bias due to lack of endoscopist blinding; relying on biopsies of the defect instead of evaluation of scars at surveillance for determining efficacy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT03462706/Prot_SAP_000.pdf